CLINICAL TRIAL: NCT01116479
Title: Randomised Feasibility Study of Optimal Transfusion Thresholds in Anaemic Cancer Patients Treated With Chemotherapy (HaemOPtimal)
Brief Title: Optimal Transfusion in Anaemic Cancer Patients Treated With Chemotherapy (HaemOPtimal)
Acronym: HaemOPtimal
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Morten Sorensen, MD, PhD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-1-2009-109
Record Dates: First submitted 2010-04-28; First posted 2010-05-05 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Cancer; Anaemia
Keywords: Anaemia, transfusion, cancer, chemotherapy, Quality of life
MeSH Terms: conditions — Neoplasms; Anemia | interventions — Blood Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Haemoglobin (<6.0 mmol/l) (Active Comparator): Blood transfusion thresholds:Haemoglobin < 6.0 mmol/l (9.9 g/dL)
  Interventions: Other: Blood transfusion
- Haemoglobin (< normal range) (Experimental): Blood transfusion threshold: Haemoglobin < 7.1 mmol/l (11.7 g/dL) for female and 8.1 mmol/l (13.4 g/dL) for males
  Interventions: Other: Blood transfusion

INTERVENTIONS:
Other: Blood transfusion — Blood transfusion with packed erythrocytes

SUMMARY:
This an open two-arm interventional randomised feasibility study in anaemic patients treated with chemotherapy. Randomisation is performed between two transfusion thresholds: Haemoglobin < 6.0 mmol/l (9.9 g/dL) versus haemoglobin < 7.1 mmol/l (11.7 g/dL) for female and 8.1 mmol/l (13.4 g/dL) for males.Primary end-point is quality of life

DETAILED DESCRIPTION:
Title:

Randomised Feasibility Study of Optimal Transfusion Thresholds in Anaemic Cancer Patients Treated with Chemotherapy (HaemOPtimal)

Background:

Cancer patients treated with chemotherapy very often become anaemic, which have profound negative impact of their quality of life. Blood transfusions can ameliorate symptoms caused by anaemia. Data are lagging with regard to what threshold should be used when offering blood transfusion.

Aim:

The primary aim is to determine which end-points reflect symptoms caused by anaemia in cancer patients treated with chemotherapy. The secondary aims are to collect data to estimate sample size in a future definitive study and to compare symptom relief using to different transfusion thresholds.

End-points:

* Numeric Rating Scale measuring fatigue, dizziness, palpitations, headache, and dyspnea.
* FACT-G,
* FACT-An (Total anemia scale) including a fatigue subscale
* Patient-assessed WHO performance status

Design:

Open two-arm interventional randomised feasibility study

Intervention:

* Blood transfusion.
* Randomisation between two transfusion thresholds:

Haemoglobin < 6.0 mmol/l (9.9 g/dL) versus Haemoglobin < 7.1 mmol/l (11.7 g/dL) for female and 8.1 mmol/l (13.4 g/dL) for males.

Population:

Cancer patients treated with chemotherapy

Inclusion criteria:

* Documented cancer
* Planned treatment with chemotherapy
* Age 18 years or older
* Informed consent

Exclusion criteria:

* Heart failure (NYHA 3 and 4)
* Prior serious complications to blood transfusion
* Medical conditions that require special considerations for blood transfusion
* Treatment with erythropoiesis-stimulating agents.

Number of patients:

Transfusion of at least 30 patients in each intervention arm. An estimated number of 90 patients will be randomised in each arm (180 in total) as a third of included patients are expected to require transfusion.

ELIGIBILITY:
Inclusion Criteria:

* Documented cancer
* Planned treatment with chemotherapy
* Age older than 18 years
* Informed consent

Exclusion Criteria:

* Heart failure (NYHA 3 and 4)
* Prior serious complications to blood transfusion
* Medical conditions that require special considerations for blood transfusion
* Treatment with erythropoiesis-stimulating agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2010-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
FACT-G, FACT-An, Numeric Rating Scale on symptoms of anaemia, Performance status | Before each cylces of chemotherapy in up to six months, and before transfusion, and daily in seven days after transfusion
  Patient assessed FACT-G (Functional Assessment of Therapy in General), FACT-An (Functional Assessment of Therapy in Anaemia), Numeric Rating Scale on symptoms of anaemia (fatigue, dizziness, dyspnea, palpitations, headache) and performance status before each cycle of chemotherapy, before transfusion and daily in seven days after transfusion

SECONDARY OUTCOMES:
Safety and transfusion complications | during or after transfusion
  Frequency of complications to blood transfusion (need for termination of transfusion due to complications, chills, fever, hives, drop in blood pressure, dyspnea, other)

CONTACTS AND LOCATIONS:
Overall Officials: Morten Sorensen, MD, Phd, Principal Investigator — Dept. of Oncology, Righospitalet, Denmark
Locations (2):
- Denmark (2):
  - Blood bank, Righospitalet, Copenhagen
  - Dept. of Oncology, Rigshospitalet, Copenhagen

REFERENCES:
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Fergusson DA, Pagano MB, Roubinian NH, Turgeon AF, Valentine S, Trivella M, Doree C, Hebert PC. Transfusion thresholds and other strategies for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2025 Oct 20;10(10):CD002042. doi: 10.1002/14651858.CD002042.pub6. PMID 41114449
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Trivella M, Roubinian N, Fergusson DA, Triulzi D, Doree C, Hebert PC. Transfusion thresholds for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2021 Dec 21;12(12):CD002042. doi: 10.1002/14651858.CD002042.pub5. PMID 34932836